## Statistical Analysis Plan

We will be looking at changes in outcomes from before to after the MBSR intervention in (a) the MBSR compared to TAU participants, and (b) within the MBSR participants. We will focus on within-persons mean differences using paired samples t-tests within the intervention group. To determine the impact of MBSR on the postoperative TKA outcomes, we will conduct multivariate analyses of variance of conceptually linked dependent variables (i.e. pain variables, mental health variables) with significant results followed up by Tukey post-hoc tests.